CLINICAL TRIAL: NCT00487487
Title: Study of Mental Fatigue in Polio Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Other Study IDs: USUHS-G192EI
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Last update posted 2007-06-18 (Estimated); Status verified 2007-03

CONDITIONS: Post-Poliomyelitis Syndrome
Keywords: Candidates for this study are survivors of paralytic poliomyelitis
MeSH Terms: conditions — Postpoliomyelitis Syndrome

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Post-Poliomyelitis Syndrome (PPS) is the term describing the new problems affecting polio survivors many years after recovery from paralytic polio. Among the symptoms, fatigue is one of the most frequent and debilitating. In addition to physical incapacitation, the fatigue of PPS also affects mental function. The term "brain fatigue" is usually used by patients to express problems on the areas of attention, concentration, memory and clear thinking. Unfortunately, little is known about cognitive fatigue of PPS patients. This study is meant to examine if mental impairment is present in PPS patients and, if so, how it interferes on the self-function of patients. Patients will undergo an interview, clinical and neurological evaluation, and a battery of screening laboratory tests to make sure they are eligible for the study. Patients who qualify will undergo neuropsychometric tests in order to assay performance in the main areas of cognitive functioning. Through this organized approach we expect to be able to determine if mental fatigue is a significant problem affecting polio survivors, what areas are most affected, and how it may interfere with daily living.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Be a survivor of poliomyelitis
* Willing to attend two clinic visits for completion of screening procedures and required tests

Exclusion Criteria:

* Suffer from medical conditions that can interfere with cognitive function, including stroke, traumatic brain injury, dementia (progressive memory loss), severe depression, psychosis or other psychiatric disorders, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Postpolio Syndrome Outpatient Research Office, Rockville, Maryland, United States